CLINICAL TRIAL: NCT02864745
Title: Functional Electrical Stimulation-assisted Cycle Ergometry in Critically Ill: Linking Deranged Muscle Physiology to Long-term Functional Outcome
Brief Title: Early Mobilization and Intensive Rehabilitation in the Critically Ill
Acronym: EMIR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Faculty Hospital Kralovske Vinohrady (Other Government)
Responsible Party: Principal Investigator, Frantisek Duska, Head of Dept. of Anaesthesia and Intensive Care, 3rd Faculty of Medicine, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-28663A
Record Dates: First submitted 2016-05-06; First posted 2016-08-12 (Estimated); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Critical Illness
Keywords: early rehabilitation; critically ill; muscle weakness; neuromuscular stimulation; functional electrical stimulation-assisted cycle ergometry; ICUAW
MeSH Terms: conditions — Critical Illness; Muscle Weakness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early rehabilitation arm (Experimental): These patients will receive very early (<48 hours after ICU admission), protocolised, intensive rehabilitation, which will include functional electrical stimulation-assisted cycle ergometry.
  Interventions: Device: functional electrical stimulation-assisted cycle ergometry
- Standard-of-care (Active Comparator): These patients will receive standard rehabilitation delivered by non-study physiotherapist.
  Interventions: Other: standard rehabilitation

INTERVENTIONS:
Device: functional electrical stimulation-assisted cycle ergometry — Early intensive rehabilitation protocol, which includes the use of functional electrical stimulation-assisted cycle ergometry
  Arms: Early rehabilitation arm
Other: standard rehabilitation — This group will receive standard rehabilitation, which will be monitored, but not protocolised.
  Arms: Standard-of-care

SUMMARY:
ICU acquired weakness contributes (ICUAW) to poor functional outcome in survivors of critical care. Most damage occurs during the first week of critical illness when patients are unable to cooperate with conventional active rehabilitation. Functional electrical stimulation-assisted cycle ergometry (FES-CE) may improve muscle function and long-term outcome. Methods: Assessor-blinded pragmatic single-centre randomized controlled trial. Adults (n=150) mechanically ventilated for < 48 hours from 4 ICUs who are estimated to need >7 days of critical care will be randomized to receive either FES-CE-based intensified rehabilitation or routine care, which will continue until ICU discharge. Primary outcome: Quality of life as measured by SF-36 score at 6 months. Secondary outcomes: functional performance at ICU discharge, cross sectional muscle diameter and nitrogen balance, and muscle power. In a subgroup we will assess insulin sensitivity and perform skeletal muscle biopsies to look at mitochondrial function, fibre typing and regulatory protein expression in response to FES-CE.

DETAILED DESCRIPTION:
Background. Functional disability, a natural consequence of weakness, is a frequent and long-lasting complication in survivors of critical illness. Over recent decades, mortality from acute critical illness has decreased with a consequent increasing number of ICU survivors. Understanding the post-ICU morbidity experienced by these survivors has become increasingly important. The greatest burdens that survivors of critical illness face are related to neuromuscular dysfunction and neuropsychological maladjustment. In particular, neuromuscular abnormalities during critical illness are common, with a median prevalence of 57%. In both patients with chronic critical illness and survivors of severe critical illness, neuromuscular weakness may be substantial and persistent, resulting in important decrements in physical function and quality of life for years after discharge. In the past, routine features of general care provided in the ICU included liberal use of sedation and immobilization of the patient, which were thought to be necessary for facilitating interventions to normalise physiological function by artificial means. Recently, there has been a paradigm shift away from this approach towards a more conservative treatment philosophy for patients in the ICU. This paradigm shift is consistent with the observation that long-term physical problems in survivors of critical illness, particularly those with respiratory failure, may result from the protracted ICU stay and period of immobilization during which the patient is receiving organ support that is essential for survival. In line, daily interruption of sedation policy has been widely adopted and proven to be beneficial and early mobilization culture is spreading quickly across ICUs. Indeed, these strategies, together with early physical therapy are the only safe and effective interventions in the prevention of long-term neuromuscular disability in survivors of intensive care. It should be stressed that in these studies, early rehabilitation is defined as starting between day 2-5 of ICU stay or as an activity beginning before ICU discharge. Standard early rehabilitation cannot be started early enough, and functional electrical stimulation-assisted cycle ergometry may be a solution to this dilemma.The first week on the ICU is critical as muscle mass and function is lost quickly. Immobility-associated muscle loss is evident as early as within18-48 hours of onset of acute critical illness or severe injury and is greatest during the first 2 to 3 weeks of critical illness. Up to 40% loss of muscle strength can occur within the first week of immobilization, with a daily rate of strength loss between 1.0% and 5.5% A 10-14% decrease in cross-sectional measurements of the rectus femoris muscle has been observed within the first week of ICU stay. Conventional rehabilitation during the first few days in the ICU is indeed limited in patients who are sedated and mechanically ventilated, and typically consists of passive limb movements, with or without the use of stretch reflex provided the earliest (within 48 hours of intubation) and largest dose of rehabilitation (26±14 min a day for patients on mechanical ventilation) and reported improvements of physical function at hospital discharge, but no measurements beyond. Active rehabilitation is delayed until the neurological condition of the patient improves enough to facilitate participation. In the sickest patients, who are at particular risk of developing ICUAW, sedation and immobility may be prolonged well beyond first week, when established damage to the muscle has already occurred. In order to achieve maximum efficacy, passive cycling and neuromuscular electrical stimulation (NMES) can be delivered simultaneously and synchronised to produce a coordinated pattern of movements. The technique is called FES-CE (functional electrical stimulation-assisted cycle ergometry). There is a large body of experience with these methods in the rehabilitation of patients with stroke and spinal cord injuries. The method is effective in preventing the loss of muscle mass and has been shown to improve anabolic resistance and insulin sensitivity in quadriplegic patients. In critical illness, pilot studies have shown NMES itself (without synchronization and the use of bicycle) to be safe, feasible and effective in maintaining muscle strength and mass. The only study of FES-CE in critically illness is the pilot trial of Parry et al., where the feasibility and safety of FES-CE was demonstrated in a small cohort of critically ill patients (8 patients received the FES-CE intervention, versus 8 controls). Patients in the intervention group showed significant improvements in the Physical Function in Intensive Care Test and a faster recovery of functional milestones (e.g. time to stand from lying, and walking on the spot).

Hypotheses H1: As most of the damage to the structure and function of skeletal muscle occurs during the first week, intensified rehabilitation, which includes FES-CE and starts within 48 hours after ICU admission, improves functional outcome of ICU survivors at 6 months when compared to the routine standard of care. H2: Intensified early rehabilitation compared to routine standard of care, shall preserve muscle mass and improve muscle power at ICU discharge. H3:Intensified early rehabilitation compared to routine standard of care shall increase insulin-mediated whole-body oxidative glucose disposal and mitochondrial functional indices. Sample size calculation:In studies of critical illness outcome at 6-months using 36-Item Short Form Health Survey (SF-36) scores, the standard deviation varied between 10-13 points. In order to have 80% power to detect 5 point difference in SF-36 score between control and intervention at the level of significance p<0.05 in the population with standard deviation (SD) of 13, we would need 108 subjects (54 in each arm). In order to allow for deaths and dropouts, the plan is to randomize 150 subjects.

Randomization. As soon as possible, but always within 48 hours of admission, participants will be randomly assigned (1:1) to receive either standard care or the intervention using offsite-independent randomization protocols (www.randomization.com). Randomization will be stratified according to presence or absence of sepsis and the availability of a biopsy at baseline. Concealed allocation will be performed using sequentially numbered opaque sealed envelopes only accessible by research personnel with no involvement in the trial.

Once consent/assent is obtained, and prior to randomisation; participants will be referred to a study physiotherapist who will administer baseline testing of muscle mass/cross-sectional area (CSA) using diagnostic ultrasound (US), and baseline blood samples will be taken Both groups will receive usual best medical and nursing care in the ICU, which include daily sedation holds when applicable and delirium management as usual in the routine practice. Respiratory physiotherapy will also be delivered without alterations. The routine standard care arm will undergo mobilisation/rehabilitation delivered by personnel not involved in the study in a usual, routine way. Details of physiotherapy treatment will be recorded but not protocolled in the standard care arm. Intervention group In the intervention arm, early rehabilitation is protocolled according to patients' condition and degree of cooperation and there will be pre-defined safety criteria, which are in accordance with current recommendations for active rehabilitation of critically ill ventilated adults. Whilst the safety criteria are binding for the study physiotherapist, the rehabilitation protocol is not and the delivery of physical exercise can be altered according to actual patient's condition. However, any alteration and the reason for it will be recorded. The intervention will start as soon as possible and always within 48 h of ICU admission, continuing until ICU discharge. Supine cycling will be delivered as per protocol on supine cycloergometer attached to a neuromuscular stimulator Surface electrodes will be applied to the gluteal, hamstrings, quadriceps and calf muscles on both legs. The intensity of muscle stimulation will be delivered at a level able to cause visible contractions (confirmed by palpation if uncertain) in all muscle groups without causing undue pain or discomfort to the participant, according to a regime specified by Parry, 2012. Once the patient is more alert, and able to participate, they will be provided with standardized encouragement to engage in therapy. To increase the intervention workload, resistance will be increased incrementally and cycling cadence. If a participant is readmitted to intensive care, the intervention will be re-initiated.

Study Procedures The ICUs are paperless and fully computerized, so vital functions and other physiological parameters are monitored and data is routinely stored to secure hospital data bases via a protected dedicated network. This includes data about nutritional intake and urinary output. Urine samples will be collected daily, surfaced with toluene and stored in a deep freeze facility for later determination of nitrogen content and 3-methyl histidine levels (to calculate muscle catabolism rate and nitrogen balance). In addition, all study patients will undergo an assessment by a study physiotherapist, which includes a measurement of rectus muscle cross-sectional area on both legs and whenever the patient regains consciousness, also muscle power by Medical Research Concil (MRC) score (standardized testing of muscle power [0-5] on 12 muscle groups on all 4 limbs, giving the score 0-60 (60 suggesting normal muscle power). Blood will be taken, plasma separated and frozen at -80 C for later analysis of cytokines and hormone levels. This assessment will be repeated at 7-day intervals and at ICU discharge. At ICU discharge, the patients and relatives will be asked to provide contact details for follow up. After 6 months, the patient or family will be contacted for structured interview as required for SF-36 questionnaire, and collected using Research and Development Organization (RAND) methodology. Whilst participants and intervention physiotherapist cannot be blinded to group allocation, research staff assessing outcome will be from separate clinical departments and thus remain blinded to treatment allocation.

Complementary Studies: Insulin resistance and mitochondrial function These studies will be performed in addition to other study procedures in a subgroup of patients, who give specific consent to it. First measurement will be performed at baseline prior to randomization, ideally the next morning after admission. Second measurement on day 7 of ICU stay, i.e. after at least 5 days of intervention. Muscle biopsy. Will be performed from vastus lateralis muscle by needle biopsy technique. The sample will be separated into three parts (50-100mg each). One part will be immediately frozen in liquid nitrogen for analysis of protein/DNA ratio and protein expression studies. The second part will be frozen in liquid nitrogen-cooled isopentane for muscle fibre typing and immunohistochemistry analysis. The third part put into culture media on ice for the preparation of homogenates and measurement of citrate-synthase activity, spectrophotometric analysis of the activity of respiratory complexes I-IV and western blot analysis of respiratory complexes. In the fresh muscle homogenates, the investigators will use high-resolution respirometry to determine the function of individual respiratory complexes in the cytosolic context and measure basic functional metabolic indices. the investigators will specifically look at the degree of mitochondrial uncoupling, respiratory chain capacity and the function of individual complexes, including glycerol-3-phosphate shuttle. Frozen muscle samples will be stored at deeply frozen for analysis of DNA/protein ratio, messenger ribonucleic acid (mRNA) and proteins involved in the regulation of proteolysis, substrate oxidation and anabolic pathways of skeletal muscle as well as immunohistochemistry and typing of muscle fibres. In addition, the investigators will look at the change of these indices after seven days of critical illness and the influence of the intervention vs. standard of care. the investigators will look at correlation of these parameters with muscle power (i.e. compare bioenergetics profile of skeletal muscle in those who develop ICUAW and in those who do not) and insulin resistance. Insulin sensitivity and substrate oxidation will be measured after overnight fasting by hyperinsulinaemic euglycemic clamp.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years;
* Mechanical ventilation, or imminent need of it at presentation;
* Predicted ICU length of stay ≥7 days;

Exclusion Criteria:

* Known primary systemic neuromuscular disease or permanent neurological damage at admission
* Severe lower limb injury or amputation
* Bedridden premorbid state
* Assessed by medical staff as approaching imminent death or withdrawal of medical treatment within 24 h
* Pregnancy
* Presence of external fixator or superficial metallic implants in lower limb
* Open wounds or skin abrasions at electrode application points
* Presence of pacemaker, implanted defibrillator or other implanted electronic medical device
* Transferred from another ICU after 24 hours of consecutive mechanical ventilation
* Presence of other condition preventing the use of FES--CE or considered unsuitable for the study by a responsible medical team
* Prior participating in another functional outcome-based intervention research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-10-04 (Actual); Primary Completion 2020-03-10 (Estimated); Study Completion 2020-03-10 (Estimated)

PRIMARY OUTCOMES:
Quality of life as per 36-Item Short Health Survey (SF-36) score | at 6 months

SECONDARY OUTCOMES:
4-item Physical Fitness in Intensive Care test | at 28 days or discharge from ICU whichever occurs earlier
  functional outcome at ICU d/c
Muscle mass measured by rectus m. crosssectional area on B-mode ultrasound | at 7 day intervals up to 28th day or discharge from ICU, whichever occurs earlier
Nitrogen balance measured in g/m2 of body surface area | at 7 day intervals up to 28th day or discharge from ICU, whichever occurs earlier
  The cumulative the difference between nitrogen intake and output
Muscle power per Medical Research Council (MRC) score | at 7 day intervals up to 28th day or discharge from ICU, whichever occurs earlier
Number of ventilator-free days | at 28 days
  Number of days, out of 28 after admission, patient has NOT been supported by mechanical ventilation
Number of rehabilitation interruptions due to physiological deterioration | at 28 days or discharge from ICU whichever occurs earlier
Number of episodes of elevated intracranial pressure | at 28 days or discharge from ICU whichever occurs earlier
Number of dialysis interruptions | at 28 days or discharge from ICU whichever occurs earlier
Length of ICU stay in days | at 6 months

OTHER OUTCOMES:
Estimated cost of care in Euro per patient per hospital stay | at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Petr Waldauf, Study Director — Faculty Hospital Kralovske Vinohrady
Locations (1):
- Kralovske Vinohrady University Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
De-dentified individual patients data will be made available in a public database. Protocol has been published in Trials.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Kress JP, Hall JB. ICU-acquired weakness and recovery from critical illness. N Engl J Med. 2014 Apr 24;370(17):1626-35. doi: 10.1056/NEJMra1209390. No abstract available. PMID 24758618
- [Background] Fan E. Critical illness neuromyopathy and the role of physical therapy and rehabilitation in critically ill patients. Respir Care. 2012 Jun;57(6):933-44; discussion 944-6. doi: 10.4187/respcare.01634. PMID 22663968
- [Background] Sacanella E, Perez-Castejon JM, Nicolas JM, Masanes F, Navarro M, Castro P, Lopez-Soto A. Functional status and quality of life 12 months after discharge from a medical ICU in healthy elderly patients: a prospective observational study. Crit Care. 2011;15(2):R105. doi: 10.1186/cc10121. Epub 2011 Mar 28. PMID 21443796
- [Background] Fan E, Dowdy DW, Colantuoni E, Mendez-Tellez PA, Sevransky JE, Shanholtz C, Himmelfarb CR, Desai SV, Ciesla N, Herridge MS, Pronovost PJ, Needham DM. Physical complications in acute lung injury survivors: a two-year longitudinal prospective study. Crit Care Med. 2014 Apr;42(4):849-59. doi: 10.1097/CCM.0000000000000040. PMID 24247473
- [Background] Herridge MS, Tansey CM, Matte A, Tomlinson G, Diaz-Granados N, Cooper A, Guest CB, Mazer CD, Mehta S, Stewart TE, Kudlow P, Cook D, Slutsky AS, Cheung AM; Canadian Critical Care Trials Group. Functional disability 5 years after acute respiratory distress syndrome. N Engl J Med. 2011 Apr 7;364(14):1293-304. doi: 10.1056/NEJMoa1011802. PMID 21470008
- [Background] Herridge MS. Mobile, awake and critically ill. CMAJ. 2008 Mar 11;178(6):725-6. doi: 10.1503/cmaj.080178. No abstract available. PMID 18332388
- [Background] Needham DM. Mobilizing patients in the intensive care unit: improving neuromuscular weakness and physical function. JAMA. 2008 Oct 8;300(14):1685-90. doi: 10.1001/jama.300.14.1685. PMID 18840842
- [Background] Slutsky AS. Neuromuscular blocking agents in ARDS. N Engl J Med. 2010 Sep 16;363(12):1176-80. doi: 10.1056/NEJMe1007136. No abstract available. PMID 20843254
- [Background] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Background] Levine S, Nguyen T, Taylor N, Friscia ME, Budak MT, Rothenberg P, Zhu J, Sachdeva R, Sonnad S, Kaiser LR, Rubinstein NA, Powers SK, Shrager JB. Rapid disuse atrophy of diaphragm fibers in mechanically ventilated humans. N Engl J Med. 2008 Mar 27;358(13):1327-35. doi: 10.1056/NEJMoa070447. PMID 18367735
- [Background] Hermans G, De Jonghe B, Bruyninckx F, Van den Berghe G. Clinical review: Critical illness polyneuropathy and myopathy. Crit Care. 2008;12(6):238. doi: 10.1186/cc7100. Epub 2008 Nov 25. PMID 19040777
- [Background] Parry SM, Berney S, Koopman R, Bryant A, El-Ansary D, Puthucheary Z, Hart N, Warrillow S, Denehy L. Early rehabilitation in critical care (eRiCC): functional electrical stimulation with cycling protocol for a randomised controlled trial. BMJ Open. 2012 Sep 13;2(5):e001891. doi: 10.1136/bmjopen-2012-001891. Print 2012. PMID 22983782
- [Background] Parry SM, Berney S, Warrillow S, El-Ansary D, Bryant AL, Hart N, Puthucheary Z, Koopman R, Denehy L. Functional electrical stimulation with cycling in the critically ill: a pilot case-matched control study. J Crit Care. 2014 Aug;29(4):695.e1-7. doi: 10.1016/j.jcrc.2014.03.017. Epub 2014 Mar 26. PMID 24768534
- [Background] Schweickert WD, Pohlman MC, Pohlman AS, Nigos C, Pawlik AJ, Esbrook CL, Spears L, Miller M, Franczyk M, Deprizio D, Schmidt GA, Bowman A, Barr R, McCallister KE, Hall JB, Kress JP. Early physical and occupational therapy in mechanically ventilated, critically ill patients: a randomised controlled trial. Lancet. 2009 May 30;373(9678):1874-82. doi: 10.1016/S0140-6736(09)60658-9. Epub 2009 May 14. PMID 19446324
- [Background] Burtin C, Clerckx B, Robbeets C, Ferdinande P, Langer D, Troosters T, Hermans G, Decramer M, Gosselink R. Early exercise in critically ill patients enhances short-term functional recovery. Crit Care Med. 2009 Sep;37(9):2499-505. doi: 10.1097/CCM.0b013e3181a38937. PMID 19623052
- [Derived] Waldauf P, Hruskova N, Blahutova B, Gojda J, Urban T, Krajcova A, Fric M, Jiroutkova K, Rasova K, Duska F. Functional electrical stimulation-assisted cycle ergometry-based progressive mobility programme for mechanically ventilated patients: randomised controlled trial with 6 months follow-up. Thorax. 2021 Jul;76(7):664-671. doi: 10.1136/thoraxjnl-2020-215755. Epub 2021 Apr 30. PMID 33931570
- [Derived] Waldauf P, Gojda J, Urban T, Hruskova N, Blahutova B, Hejnova M, Jiroutkova K, Fric M, Jansky P, Kukulova J, Stephens F, Rasova K, Duska F. Functional electrical stimulation-assisted cycle ergometry in the critically ill: protocol for a randomized controlled trial. Trials. 2019 Dec 16;20(1):724. doi: 10.1186/s13063-019-3745-1. PMID 31842936